CLINICAL TRIAL: NCT02641990
Title: A Phase 1, Randomized, Double-blind, Placebo-Controlled, Crossover Study to Assess the Effect of ITCA 650 on the Pharmacokinetics and Pharmacodynamics of a Combination Oral Contraceptive in Healthy Premenopausal Female Subjects
Brief Title: Study of the Effect of ITCA 650 on the PK/PD of Oral Contraceptive in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Intarcia Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: ITCA 650-CLP-116
Record Dates: First submitted 2015-12-18; First posted 2015-12-30 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2016-03

CONDITIONS: Healthy Adult Premenopausal Female Volunteers
MeSH Terms: interventions — Exenatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): ITCA 650 20/60 mcg/day, ITCA placebo
  Interventions: Drug: ITCA 650 20/60 mcg/day, ITCA placebo
- Group 2 (Experimental): ITCA placebo, ITCA 650 20/60 mcg/day
  Interventions: Drug: ITCA placebo, ITCA 650 20/60 mcg/day

INTERVENTIONS:
Drug: ITCA 650 20/60 mcg/day, ITCA placebo — ITCA 650 osmotic mini pump delivering exenatide 20/60 mcg/day and Levora® for 28 days, followed by ITCA osmotic mini pump delivering placebo and Levora® for 28 days
  Arms: Group 1
Drug: ITCA placebo, ITCA 650 20/60 mcg/day — ITCA osmotic mini pump delivering placebo and Levora® for 28 days, followed by Levora® and ITCA 650 osmotic mini pump delivering exenatide 20/60 mcg/day and Levora® for 28 days
  Arms: Group 2

SUMMARY:
A Phase 1, randomized, double-blind, placebo-controlled, crossover study to assess the effect of ITCA 650 on the pharmacokinetics (PK) of once daily administration of Levora® (ethinyl estradiol 0.3 mg (EE) and levonorgestrel 0.15 mg (LNG) in healthy premenopausal female subjects.

ELIGIBILITY:
Inclusion Criteria:

* Women of childbearing potential.
* Use of a combination oral contraceptive ≥3 months immediately prior to screening.
* Willing to use an additional adequate method of contraception during the study and until 1 additional menstrual cycle following the end-of-study (EOS) visit. Adequate methods of contraception for women of child bearing potential (WOCBP) include: mechanical products (ie, intrauterine device [IUD]-copper IUD); or barrier methods (eg, diaphragm, condoms, cervical cap) with spermicide.
* Body mass index (BMI) ≥19 and ≤32 kg per meter squared.
* Weight ≥50 and ≤100 kg.
* Non-smoker or ex-smoker for >6 months prior to screening (and has stopped using other nicotine products ≥2 weeks prior to screening).

Exclusion Criteria:

* History of type 1 or type 2 diabetes.
* Received implanted contraceptives within 6 months prior to screening or injected contraceptives within 12 months prior to screening.
* History or evidence, within the last 6 months prior to the Screening Visit, of myocardial infarction, coronary revascularization (coronary artery bypass grafting or percutaneous coronary intervention), unstable angina, or cerebrovascular accident or stroke.
* History of uncontrolled hypertension.
* History or evidence of acute or chronic pancreatitis.
* History of liver disease.
* History of medullary thyroid cancer or a personal or family history of multiple endocrine neoplasia type 2.
* Poor thyroid, liver, or renal function.
* Weight loss surgery or requires weight loss medications.
* History of malignancy (not including basal or squamous cell carcinoma of the skin with past 5 years). (Subjects who have been disease free for 5 years may be included.)
* Estrogen-dependent growths; undiagnosed vaginal bleeding.
* History of active alcohol or substance abuse.
* Regular daily consumption of more than 12 g of alcohol in any form.
* Excessive in xanthine consumption (more than 5 cups of coffee or equivalent per day).
* Treatment with medications that affect GI motility.
* Any condition that would affect drug transit time or absorption (eg, gastrointestinal bypass surgery, partial or total gastrectomy, small bowel resection, chronic diarrhea, vagotomy, chronic gastroesophageal reflux disease, malabsorption, colostomy, Crohn's disease, ulcerative colitis, or celiac sprue).
* History of hypersensitivity to exenatide.
* Contraindications or warnings according to the specific label(s) for EE and/or LNG therapy.
* Women that are pregnant, lactating, or planning to become pregnant.
* Any use of anticoagulants with the exception of those given in prophylaxis prior to surgical intervention.
* History of or positive results on screening tests for hepatitis B and/or hepatitis C and/or human immunodeficiency virus (HIV).
* Recent surgery or planned in-patient surgery, dental procedure, or hospitalization during the study.
* History of migraine if aged >35 years or has focal symptoms associated with migraine.
* History of thrombophlebitis, thromboembolic disorders, or deep vein thrombophlebitis.
* Fasting triglycerides above upper limit of normal at Screening.
* Any gastrointestinal complaints within 7 days prior to first dosing.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2015-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration-time curve at steady state (AUCss) for ethinyl estradiol and levonorgestrel | from baseline to 13 weeks
Maximum steady state plasma concentration (Cmax,ss) for ethinyl estradiol and levonorgestrel | from baseline to 13 weeks

SECONDARY OUTCOMES:
Time to maximum steady state plasma concentration (tmax,ss) for ethinyl estradiol and levonorgestrel | baseline to 13 weeks
  Immunogenicity parameters:
  - ADA (anti-exenatide antibodies)
  Safety parameters:
  - Treatment-emergent AEs (TEAEs) including any events local to the placement site, clinical laboratory measurements, ECGs, vital signs and physical examinations.
Apparent plasma clearance at steady-state (CL/Fss) for ethinyl estradiol and levonorgestrel | baseline to 13 weeks

OTHER OUTCOMES:
Additional Outcome Measure 1 | 13 weeks
  Pharmacodynamics - FSH
Additional Outcome Measure 2 | 13 weeks
  Pharmacodynamics - LH
Additional Outcome Measure 3 | 13 weeks
  Pharmacodynamics - progesterone

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - QPS/Miami Research Associates, Miami, Florida
  - Compass Research, Orlando, Florida

IPD SHARING:
Plan to Share IPD: No